CLINICAL TRIAL: NCT03140579
Title: Estimation of Long Term PEEP Effect on Lung Homogeneity and Recruitment Using APRV Ventilation:Measurement of End Expiratory Lung Volume With Nitrogen Wash-out/wash-in Technique and End Expiratory Lung Impedance With EIT at Different Times.
Brief Title: Effect of PEEP on Lung Recruitment and Homogeneity Over Time in Moderate to Severe ARDS
Acronym: APRV
Status: Withdrawn | Type: Observational
Why Stopped: Study not undertaken due to COVID and capacity
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 123456789
Record Dates: First submitted 2017-05-02; First posted 2017-05-04 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: ARDS; Critical Illness; Ventilator-Induced Lung Injury
Keywords: recruitment; lung homogeneity; airway pressure release ventilation
MeSH Terms: conditions — Critical Illness; Ventilator-Induced Lung Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: APRV — Airway pressure release ventilation is a method of inverse ventilation, where high levels of positive end expiratory pressure are maintained to optimise oxygenation with brief releases of pressure to allow ventilation and release carbon dioxide. It is an approved and frequently used method of ventilation.

SUMMARY:
This study evaluates the effect of airway pressure release ventilation (APRV) on lung homogeneity and recruitment in patients with moderate to severe acute respiratory distress syndrome (ARDS).

It will do this by comparing the homogeneity of ventilation and recruitment prior to a patient being ventilated on APRV, and at 30, 60 and 120 minutes after starting APRV.

DETAILED DESCRIPTION:
Ventilator-induced lung injury (VILI) is a well-recognised problem of ventilation in patients with ARDS, and is currently treated with lung-protective ventilation, which limits tidal volumes and airway pressures by applying higher levels of positive-end expiratory pressure (PEEP). However, it is not known whether higher levels of PEEP increases recruitment and homogeneity of ventilation within the lungs.

APRV is a mode of inverse ventilation, where high levels of PEEP are maintained with brief releases of pressure, and has been proposed as an appropriate method of ventilation in patients with ARDS.

This study will assess homogeneity of ventilation and recruitment in 15 patients before APRV is started, and 30, 60 and 120 mins after commencing APRV. It will do this using Electrical Impedance Tomography (EIT), nitrogen wash in/wash out technique, and lung strain.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and < 80 years

  * Weight > 35 Kg and BMI < 40
  * Informed consent according to local regulations
  * Hemoglobin ≥ 70 g/dl
  * Haemodynamically stable > 4 hours
  * Moderate to severe ARDS (PaO2/FIO2 < 26.6 kPa with positive end-expiratory pressure (PEEP) > 5 cmH2O) as per Berlin definition of ARDS

Exclusion Criteria:

* Expected survival < 72 hours

  * Suspected pregnancy (negative pregnancy test required for women of child-bearing potential)
  * Open abdomen
  * Documented or suspected raised intracranial pressure
  * Active air leak (pneumothorax, pneumomediastinum, subcutaneous emphysema)
  * Morbid obesity BMI > 40
  * Recent < 1 week cardiac or thoracic surgery
  * Unstable thorax and sternum with paradoxical chest wall movement
  * Severe Chronic Respiratory Disease (COPD) - GOLD 3 or 4 emphysema with bullae
  * Severe smoking (> 40 pack-year history)
  * Liver Failure: Child-Pugh Class C
  * Massive ascites
  * Lung fibrosis
  * Severe cardiac disease (one of the following): New York Heart Association Class III or IV, acute coronary syndrome or persistent ventricular tachyarrhythmias
  * Sickle cell disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All Patients admitted to ICU ventilated with moderate or severe ARDS, based on the Berlin definition of ARDS.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-06-01 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
To compare lung homogeneity estimated with EIT upon commencing APRV (APRVpre) and after 30 - 60 - 120 min of APRV ventilation (APRV30, APRV60, APRV120) in patients with moderate to severe ARDS | 30, 60 and 120 mins
  EIT will be measured at time APRVpre during a "low-flow maneuver" consisting of a brief switch to PC ventilation: with a flow of 4 L/min, airway pressure will be gradually increased up to 30 cmH20 in order to see how the lung changes elastically minimising resistance. EIT will also be measured after 30 min (time APRV30), 60 min (time APRV60), 120 min (time APRV120) since APRV has started.

SECONDARY OUTCOMES:
To assess recruitment at the beginning and after the end of APRV ventilation in patients with moderate-severe ARDS. | 2 hours
  To assess recruitment measuring change in end expiratory lung impedance (EELI) with EIT technique, and EELV with nitrogen wash-out/wash-in technique.
To compare lung strain measured at APRVpre and after the end of APRV ventilation (APRVpost) in patients with moderate-severe ARDS | 2 hours
  Strain will be calculated at time APRVpre using the strain formula (TV/EELV)

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Camporota, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guys and St Thomas NHS Foundation, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
All shared data will be as a mean and not as individual